CLINICAL TRIAL: NCT00650962
Title: Does Longer Pre-shock Cardiopulmonary Resuscitation Improve the Outcome of Patients With Out-of-hospital Cardiac Arrest? A Randomized Control Trial.
Brief Title: Pre-shock Cardiopulmonary Resuscitation to Patients With Out-of-hospital Resuscitation, A Randomised Clinical Trial
Acronym: CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200710019R; NSC 962314B002018
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-12

CONDITIONS: Cardiac Arrest
Keywords: CPR; Preshock CPR; OHCA; EMS
MeSH Terms: conditions — Heart Arrest | interventions — Cardiopulmonary Resuscitation; Defibrillators

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPR first (Active Comparator): Compression First (CF)
  Interventions: Other: cardiopulmonary resuscitation
- Analysis First (Active Comparator): Rhythm analysis first
  Interventions: Other: Rhythm analysis

INTERVENTIONS:
Other: cardiopulmonary resuscitation — 10 cycles of 30:2 cardiopulmonary resuscitation before rhythm analysis by AED
  Other Names: automatic external defibrillator
  Arms: CPR first
Other: Rhythm analysis — Rhythm analysis as soon as AED is ready
  Other Names: cardiopulmonary resuscitation; automatic external defibrillator
  Arms: Analysis First

SUMMARY:
1. Pre-shock cardiopulmonary resuscitation might benefit the survival of out-of-hospital cardiac patients with ventricular fibrillation / ventricular tachycardia in a post-hoc analysis of a prehospital trial conducted in Europe (L.Wik,2002). However, it's effectiveness in the Asian countries, where most firstly recorded rhythm in out-of-hospital cardiac arrests patients were asystole/pulseless electric activity rather than ventricular fibrillation / ventricular tachycardia, were not explored yet.
2. This trial was designed to exam if pre-shock cardiopulmonary resuscitation by emergency medical technicians improves the outcome of all out-of-hospital cardiac arrest patients in an Asian metropolitan city.

DETAILED DESCRIPTION:
1. Different from data from the Western countries, non-shockable rhythm (Asystole/pulseless electric activity) was responsible for most out-of-hospital cardiac arrest patients(80%~90%) in metropolitan Taipei.
2. Response time in Taipei emergency medical service was longer than 5 minutes.
3. Bystander cardiopulmonary resuscitation rate were relatively low in Taipei.
4. Cardiopulmonary resuscitation is the only known method to save out-of-hospital cardiac arrest patients with asystole/pulseless electric activity. For those suffered from ventricular fibrillation/ ventricular tachycardia,previous studies revealed pre-shock cardiopulmonary resuscitation may have the potential to improve the outcome.
5. Study hypothesis: Compared with current standard resuscitative sequence (basic life support protocol in Guideline 2005), longer pre-shock cardiopulmonary resuscitation provided to all out-of-hospital cardiac arrest patients in Taipei may improve the outcome of them.

ELIGIBILITY:
Inclusion Criteria:

* Patients with out-of-hospital cardiac arrest

Exclusion Criteria:

* Trauma
* Age < 18y/o
* Airway obstruction
* Submersion
* Sign of obvious death
* existing do not resuscitate (DNAR) order
* family refusal
* preceding CPR by BLS teams for longer than 2 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1666 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Sustained ROSC >= 2 hours | 180 days

SECONDARY OUTCOMES:
surival to ICU admission | 180 days
survival to hospital discharge | 180 days
Rates of good neurology recovery (CPC 1 &2) | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Huei-Ming Ma, MD, PHD, Principal Investigator — Department of Emergency Medicine, NTUH.
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan